CLINICAL TRIAL: NCT00481455
Title: A Single-Center, Open-Label, Phase II, Safety and Efficacy Study of Panzem Nanocrystal Colloidal Dispersion Administered Orally in Combination With Protracted Oral Fixed-Dose Temozolomide to Patients With Recurrent Glioblastoma Multiforme
Brief Title: Phase 2 Study of Panzem Nanocrystal Colloidal Dispersion (NCD) in Combination With Fixed-Dose Temozolomide to Patients With Recurrent Glioblastoma Multiforme (GBM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CASI Pharmaceuticals, Inc. (Industry)
Responsible Party: Chief Medical Officer, EntreMed, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ME-CLN-007
Record Dates: First submitted 2007-05-30; First posted 2007-06-01 (Estimated); Last update posted 2008-11-25 (Estimated); Status verified 2008-11

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: Glioblastoma Multiforme; temozolomide
MeSH Terms: conditions — Glioblastoma | interventions — 2-Methoxyestradiol; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Panzem NCD; Drug: Temozolomide

INTERVENTIONS:
Drug: Panzem NCD — 2000 mg q8h, continuous dosing in 28 day cycles
  Other Names: 2-methoxyestradiol; 2ME2
Drug: Temozolomide — Fixed dose

SUMMARY:
The purpose of this study is to evaluate the anti-tumor activity and safety of Panzem NCD given in combination with daily oral fixed-dose temozolomide in patients with recurrent glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

1. A histologically confirmed diagnosis of a recurrent/progressive primary WHO grade IV malignant glioma (glioblastoma multiforme or gliosarcoma). Patients with recurrent disease whose diagnostic pathology confirmed WHO grade IV malignant glioma (glioblastoma multiforme or gliosarcoma) will not need re-biopsy. Patients with prior low-grade glioma are eligible if histologic assessment demonstrates transformation to WHO grade IV malignant glioma. Pathology must be confirmed at Duke University Medical Center
2. Male or female, aged greater than or equal to 18 years.
3. An interval of at least 2 weeks between prior surgical resection (if conducted) or any major surgery or 4 weeks between prior radiotherapy or chemotherapy (except nitrosoureas which require 6 weeks) and enrollment in this protocol unless there is unequivocal evidence of tumor progression and the patient has recovered from toxicities associated with those therapies. However, patients treated with chemotherapeutic agents such as VP-16 who would normally be retreated after shorter intervals (e.g. 21 days on, 7 days off schedule) may be treated at the usual starting time even if less than 4 weeks from the last prior dose of chemotherapy.
4. Karnofsky performance score greater than or equal to 70%.
5. Hematocrit > 29%, absolute neutrophil count > 1,500 cells/*L, platelets > 100,000 cells/*L.
6. Serum creatinine < 1.5 X upper limit of normal (ULN), serum glutamic oxaloacetic transaminase < 2.5 X ULN; and bilirubin < 1.5 times ULN.
7. Signed informed consent form and authorization for use and disclosure of protected health information approved by the Institutional Review Board (IRB) prior to patient entry.
8. If sexually active, patients must use contraceptive measures for the duration of the treatments and for 4 weeks following end of study medication.

Exclusion Criteria:

1. Current, active systemic bleeding or excessive risk of bleeding as defined by the following: stroke within the previous 6 months, history of central nervous system or intraocular bleed, history of septic endocarditis or evidence of intratumor hemorrhage on pretreatment diagnostic imaging, except for stable post operative grade 1 hemorrhage.
2. Female patients who are pregnant or breastfeeding or adults of reproductive potential not employing an effective method of birth control. (Women of childbearing potential must have a negative pregnancy test within 48 hours prior to administration of study medication).
3. Concurrent severe and/or uncontrolled medical disease (i.e. uncontrolled diabetes, congestive cardiac failure, myocardial infarction within 6 months, poorly controlled hypertension, history of labile hypertension, history of poor compliance with antihypertensive regimen, chronic renal disease, or active uncontrolled infection) that could compromise participation in the study.
4. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of study medication (i.e. ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, bowel obstruction, or inability to swallow the liquid).
5. Requirement for therapy with coumadin (warfarin sodium).
6. Patient is < 1 year free of another primary malignancy except if the other primary malignancy is not currently clinically significant or requiring active intervention, or if other primary malignancy is a basal cell skin cancer or a cervical carcinoma in situ. Existence of any other malignant disease is not allowed.
7. Patients unwilling to or unable to comply with the protocol.
8. Grade 2 or greater peripheral sensory neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
6-month progression free survival and median overall survival for patients receiving at least one dose | Every 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, Principal Investigator — Duke University
Locations (1):
- The Brain Tumor Center, Duke University Medical Center, Durham, North Carolina, United States